CLINICAL TRIAL: NCT01994057
Title: Retrospective Study Based on Somatic Mutations, Genetic Polymorphisms and Metabolomics Related to Individual Variations of Drug Effect and Adverse Drug Reaction of EGFR-TKIs,Gefitinib and Erlotinib in Non-small Cell Lung Cancer Treatment.
Brief Title: A Retrospective Study of EGFR-TKIs,Gefitinib, Erlotinib and Osimertinib in NSCLC Patients Treatment
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Guan shaoxing, PHD, PHD, Sun Yat-sen University
Other Study IDs: 2012ZX09506001-004 (2); (2) (Other: China: National Natural Science Foundation)
Record Dates: First submitted 2013-11-01; First posted 2013-11-25 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC); EGFR-TKI Resistant Mutation; EGFR-TKI Sensitizing Mutation; Germline Mutations; Somatic Mutation
Keywords: Non-small cell lung cancer (NSCLC);; EGFR-TKI;; Pharmacogenetics;; Precision medicine; somatic mutations ,germline mutations;
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 1. FFPE samples of tissue needle biopsy were used for EGFR mutation detection.
  2. EDTA-whole blood was centrifuged at 4000rpm*10min,plasma was separated within four hours for somatic mutation detection.The remaining samples were used for germline mutation detection. All the blood samples were frozen in -80℃ until analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- sensitive group; resistant group: sensitive patients were defined as patients reached CR or PR after first month administration,SD after first three months administration.
  resistant patients were defined as patients reached PD after first month administration and first three months administration

SUMMARY:
For patients of advanced NSCLC (non small cell lung cancer) , Individualized cancer therapy has been widely accepted since the success of crizotinib administration based on EML4-ALK fusion gene detection and gefitinib and erlotinib administration based on EGFR-TKIs sensitive mutations.From clinical points of view ,individual differences often occur between different patients, leading diverse effect in ADR and drug effect.Meanwhile ,the drug effect and adverse drug reaction was significantly influenced by the pharmacokinetic factors and pharmacodynamic factors.In this research ,we try to establish a more sensitive method to detect sensitive mutations in plasma and discover the correlation between somatic and germline mutations , trough concentration and EGFR-TKI drug effect, the association between ADME-associated SNP ,trough concentration and EGFR-TKI adverse effect .Furthermore, in vivo and in vitro research is also crucial for rational explanation for these clinical phenomenon.

DETAILED DESCRIPTION:
The ADME-associated SNPs included are CYP3A4,CYP3A4,CYP1A1,CYP2D6, ABCB1,ABCG2 and so on .The somatic mutations included are EGFR ,K-RAS ,ALK and so on

ELIGIBILITY:
Inclusion Criteria:

The main patient entry criteria included: age≥ 18 years ; histologically and cytologically proved NSCLC; Eastern cooperative oncology group performance status (ECOG PS)≤2; adequate hematological , renal, and hepatic functions. Exclusion Criteria:

uncontrolled systemic disease ,any evidence of clinically active interstitial lung diseases, and other chemotherapy at the time of inclusion. The protocol was approved by the Ethical Committee of Cancer Center of Sun Yat-Sen University (CCSU), and written informed consent was obtained form each patient.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced or metastatic NSCLC (non-small cell lung cancer) patients; administrated with gefitinib,erlotinib .
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-09; Primary Completion 2025-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | The length of time from either the date of diagnosis to that patients diagnosed with the disease are still alive
  Excluding clinical deterioration without evidence of objective progression according to the Response Evaluation Criteria In Solid Tumors (RECIST), or death from any cause.

SECONDARY OUTCOMES:
Number of patients with objective response and adverse events | one month, three month
  Objective responses (complete response plus partial response) and disease control (objective response plus stable disease
  ≥6 weeks) were established according to RECIST.And adverse events was established according to NCI-CTC .

OTHER OUTCOMES:
Number of patients with ADR | one month, three month
  Such as rash

CONTACTS AND LOCATIONS:
Overall Officials: Min Huang, Professor, Study Chair — school of pharmaceutical sciences , SunYat-senU
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Zhang L, Ma S, Song X, Han B, Cheng Y, Huang C, Yang S, Liu X, Liu Y, Lu S, Wang J, Zhang S, Zhou C, Zhang X, Hayashi N, Wang M; INFORM investigators. Gefitinib versus placebo as maintenance therapy in patients with locally advanced or metastatic non-small-cell lung cancer (INFORM; C-TONG 0804): a multicentre, double-blind randomised phase 3 trial. Lancet Oncol. 2012 May;13(5):466-75. doi: 10.1016/S1470-2045(12)70117-1. Epub 2012 Apr 17. PMID 22512843
- [Background] Kelly K, Chansky K, Gaspar LE, Albain KS, Jett J, Ung YC, Lau DH, Crowley JJ, Gandara DR. Phase III trial of maintenance gefitinib or placebo after concurrent chemoradiotherapy and docetaxel consolidation in inoperable stage III non-small-cell lung cancer: SWOG S0023. J Clin Oncol. 2008 May 20;26(15):2450-6. doi: 10.1200/JCO.2007.14.4824. Epub 2008 Mar 31. PMID 18378568
- [Background] Fukuoka M, Yano S, Giaccone G, Tamura T, Nakagawa K, Douillard JY, Nishiwaki Y, Vansteenkiste J, Kudoh S, Rischin D, Eek R, Horai T, Noda K, Takata I, Smit E, Averbuch S, Macleod A, Feyereislova A, Dong RP, Baselga J. Multi-institutional randomized phase II trial of gefitinib for previously treated patients with advanced non-small-cell lung cancer (The IDEAL 1 Trial) [corrected]. J Clin Oncol. 2003 Jun 15;21(12):2237-46. doi: 10.1200/JCO.2003.10.038. Epub 2003 May 14. PMID 12748244
- [Background] Kris MG, Natale RB, Herbst RS, Lynch TJ Jr, Prager D, Belani CP, Schiller JH, Kelly K, Spiridonidis H, Sandler A, Albain KS, Cella D, Wolf MK, Averbuch SD, Ochs JJ, Kay AC. Efficacy of gefitinib, an inhibitor of the epidermal growth factor receptor tyrosine kinase, in symptomatic patients with non-small cell lung cancer: a randomized trial. JAMA. 2003 Oct 22;290(16):2149-58. doi: 10.1001/jama.290.16.2149. PMID 14570950
- [Background] Guan S, Chen X, Chen Y, Wan G, Su Q, Liang H, Yang Y, Fang W, Huang Y, Zhao H, Zhuang W, Liu S, Wang F, Feng W, Zhang X, Huang M, Wang X, Zhang L. FOXO3 mutation predicting gefitinib-induced hepatotoxicity in NSCLC patients through regulation of autophagy. Acta Pharm Sin B. 2022 Sep;12(9):3639-3649. doi: 10.1016/j.apsb.2022.02.006. Epub 2022 Feb 15. PMID 36176901
- [Background] Guan S, Chen X, Chen Y, Xie W, Liang H, Zhu X, Yang Y, Fang W, Huang Y, Zhao H, Zhuang W, Liu S, Huang M, Wang X, Zhang L. FOXM1 Variant Contributes to Gefitinib Resistance via Activating Wnt/beta-Catenin Signal Pathway in Patients with Non-Small Cell Lung Cancer. Clin Cancer Res. 2022 Sep 1;28(17):3770-3784. doi: 10.1158/1078-0432.CCR-22-0791. PMID 35695863
- [Derived] Guan S, Chen X, Wei Y, Wang F, Xie W, Chen Y, Liang H, Zhu X, Yang Y, Fang W, Huang Y, Zhao H, Zhang X, Liu S, Zhuang W, Huang M, Wang X, Zhang L. Germline USP36 Mutation Confers Resistance to EGFR-TKIs by Upregulating MLLT3 Expression in Patients with Non-Small Cell Lung Cancer. Clin Cancer Res. 2024 Apr 1;30(7):1382-1396. doi: 10.1158/1078-0432.CCR-23-2357. PMID 38261467
- See also: department of medical oncology ,Cancer Center ,Sun Yat-sen University — http://www.sysucc.org.cn/